CLINICAL TRIAL: NCT00699166
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter 2-Week Pilot Study to Evaluate the Efficacy, Safety and Tolerability of DNK333 (25 and 100 mg Bid) Given Orally in Female Patients With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Efficacy, Safety and Tolerability of DNK333 (25 and 100 mg Bid) in Women With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Acronym: CDNK333B2201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDNK333B2201
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Diarrhea; gastrointestinal functional disorder; IBS-D
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Gastrointestinal Diseases | interventions — DNK 333

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DNK333
- 2 (Experimental)
  Interventions: Drug: DNK333
- 3 (Placebo Comparator)
  Interventions: Drug: DNK333

INTERVENTIONS:
Drug: DNK333 — 25 mg and 100 mg oral doses, each taken twice daily

SUMMARY:
This study will evaluate the tolerability, safety and efficacy of DNK333 against diarrhea caused by Irritable Bowel Syndrome in women.

ELIGIBILITY:
Inclusion Criteria:

Women of 18 - 65 years of age with IBS-D as defined by the Rome II criteria. The Rome II criteria is a system used for diagnosing functional gastrointestinal disorders such as irritable bowel syndrome. It involves completing of a questionnaire about gastrointestinal symptoms.

Note: Patients who are 50 years of age and older must have had a colonoscopy OR a flexible sigmoidoscopy plus a double-contrast barium enema within the past 5 years, which demonstrated no clinically significant findings.

Clinically significant findings may include but are not limited to malignant tumors, multiple (≥3) or advanced adenomas, inflammatory bowel disease, diverticulitis, ischaemic colitis, lymphocytic colitis, or collagenous colitis.

Patients must report ≥ 3 days with IBS-related abdominal pain/discomfort plus at least 3 days of 2 or more of the following events during the baseline period:

1. ≥ 3 bowel movements/day
2. Bowel urgency
3. Loose or watery stool

   -

   Exclusion Criteria:
   * Patients who answer "yes" to either or both of the two weekly satisfaction questions during the baseline period. The questions are: (1) Over the past week did you have satisfactory relief of your IBS-related abdominal pain/discomfort? (2) Over the last week did you have satisfactory relief of your overall IBS-D symptoms?
   * Patients with hard or lumpy stools for more than one day during the baseline period
   * Lactose intolerant patients relieved on a lactose free diet
   * Use of antidepressants (tricyclic, SSRI etc), opioid analgesic drugs or drugs specifically affecting bowel motility during the course of the trial.
   * Women of child-bearing potential who do not use an acceptable methods of contraception
   * Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average stool form score at 2 weeks | 2 weeks

SECONDARY OUTCOMES:
Change from baseline in average score at week 1, week 2: Abdominal pain/discomfort, bloating; satisfaction with bowel habits; weekly stool frequency; percent of days with satisfactory control of bowel urgency; satisfactory relief of overall IBS symptoms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis
Locations (29):
- United States (29):
  - Anniston, Alabama
  - Huntsville, Alabama
  - Northport, Alabama
  - Tucson, Arizona
  - North Little Rock, Arkansas
  - Orange, California
  - Riverside, California
  - San Diego, California
  - Torrance, California
  - Bristol, Connecticut
  - Hartford, Connecticut
  - Hollywood, Florida
  - Indianapolis, Indiana
  - Arkansas City, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Mexico, Missouri
  - Washington, Missouri
  - Lincoln, Nebraska
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Beaver Falls, Pennsylvania
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Lake Jackson, Texas
  - Salt Lake City, Utah